CLINICAL TRIAL: NCT05008562
Title: USG evaluatıon of COVID-19 Related Muscle Mass Change in the ICU
Brief Title: How COVID-19 Effects to Muscle Mass Change ın ICU?
Status: Completed | Type: Observational
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, GUNES COMBA CEBECI, specialist, Ondokuz Mayıs University
Other Study IDs: 25-2021
Record Dates: First submitted 2021-06-11; First posted 2021-08-17 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2021-08

CONDITIONS: SARS-CoV-2 Acute Respiratory Disease; Sarcopenia; ICU Acquired Weakness; Critical Illness Myopathy
Keywords: Sarcopenia; ICU Acquired Weakness; SARS-CoV-2 Acute Respiratory Disease,
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 RELATED MUSCLE MASS CHANGE IN THE INTENSIVE CARE UNIT: Patients over the age of 18 who are hospitalized in our intensive care unit with a diagnosis of COVID-19 will be included in the study.
  The day the patients are admitted to the intensive care unit will be considered the 1st day of the study. SOFA, qSOFA, APACHE II, CRP, procalcitonin values will be recorded on the first day. On the first day of our patients, rectus femoris muscle thickness measurement will be done ultrasonographically (bilateral). In addition, bilateral thigh circumference will be measured anthropometrically (with a tape measure). It is planned to evaluate the muscle strength of the patients according to the MRC (Medical Research Council) scoring.
  In addition to these measurements, the creatine kinase values in the routine clinical follow-up of the patients, the differences between the fluid intake and output values, inotropic supplements used in their treatment, diuretic needs, and neuromuscular blocker use will also be noted.
  Interventions: Other: COVID-19 RELATED MUSCLE MASS CHANGE IN THE INTENSIVE CARE UNIT

INTERVENTIONS:
Other: COVID-19 RELATED MUSCLE MASS CHANGE IN THE INTENSIVE CARE UNIT — there is no interventions to the patients.

SUMMARY:
Critical illness myopathy and neuropathy are associated with prolonged mechanical ventilation, resulting in increased morbidity and mortality in intensive care units, .the investigators aimed to determine the decrease in muscle mass and risk factors that are important causes for the development of myopathy in COVID-19 (+) patients followed in intensive care unit. The study will also evaluate the relationships of patients withthe investigators intensive care-associated muscle weakness (ICU-AW) with other intensive care patient weight scores (SOFA, APACHE II, q SOFA).

Sensitivity of anthropometric measurements and ultrasonographic measurements will be compared in the evaluation of sarcopenia. The length of hospital stay, mechanical ventilation time, patient outcomes (mortality/morbidity) information of patients with COVID-19 pneumonia followed in the intensive care unit will be evaluated.

DETAILED DESCRIPTION:
Sarcopenia (muscle weakness) is one of the geriatric syndromes that increases in frequency with age and is characterized by a decrease in muscle mass, strength and performance. Sarcopenia that occurs with aging is called primary sarcopenia, but sarcopenia can also occur due to secondary causes such as malnutrition, chronic diseases and immobility. One of the most important risk factors is advanced age. The prevalence of sarcopenia, which has been reported between 5% and 13% in a decade, can reach up to 50% over the age of 80. Sarcopenia is an important health problem that can cause loss of mobility, risk of functional dependence, risk of falling, increase in hospital stay, and consequently increase in morbidity and mortality, especially in elderly patients.

In order to be able to say sarcopenia, the investigators need to show that there is a decrease in muscle mass and, in addition, muscle strength and/or performance. Bio-electrical impedance analysis, anthropometric measurements or radiological measurements can be used among the most commonly used methods when evaluating muscle mass. However, there is no single gold standard measurement. Cross-sectional muscle area measurements, lean mass measurements and calf circumference measurements are the most commonly used muscle mass determination methods.

Ultrasonographic measurement of the rectus femoris muscle is a muscle mass measurement technique that has been used frequently recently. The most important measurement method used as a standard for muscle strength measurement is hand grip strength. The hand grip strength values reported for weakness acquired in the intensive care unit are at lower limits. <11 kg in male patients and <7 kg in female patients are considered significant limits for ICU-AW (intensive care unit-aquire weakness). However, there are some difficulties in evaluating muscle strength in intensive care patients. Most importantly, most of the patients are bedridden, immobile, receiving ventilation support, unable to cooperate, and who will not be conscious because they are under anesthesia. Apart from this, there are some measurement methods by sending magnetic or electrophysiological stimuli to the peripheral nerves in intensive care patients for muscle strength measurement, but they are mostly applied for clinical studies for now, due to the fact that they are invasive measurement methods and there are not enough equipped centers to apply them. In conclusion, sufficient number of studies examining this issue are required to reach a consensus on how to diagnose sarcopenia in intensive care patients.

In today's conditions, patients with a diagnosis of COVID-19 pneumonia are followed in the majority of intensive care units. In the study, patients with a diagnosis of COVID-19 followed in the intensive care unit will be evaluated. It is aimed to monitor, detect and investigate the factors affecting the muscle weakness of the disease, which the investigatorshave just met during the pandemic the investigators are in, and which causes different systemic involvement. There is no previous study on this subject in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Being in the Intensive Care Unit

  * Over the age of 18
  * Diagnosed with COVID-19 pneumonia

Exclusion Criteria:

* Under the age of 18

  * Pregnancy
  * Having a cardiac pacemaker
  * Amputated lower limbs Having severe venous insufficiency or major injuries to their lower extremities
  * Having neuromuscular disease
  * Malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Being in the Intensive Care Unit
  * Over the age of 18
  * Diagnosed with COVID-19 pneumonia
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Effects of COVID-19 ARDS on ICU-AW development, anthropometric measurement, | Change from baseline in thigh circumference at 21 days
  The measurements of the patients were recorded as anthropometric ( thigh circumference) on the 1st, 7th, 14th and 21st days. Thigh circumference (centimeter) was measured anthropometrically with a tape measure (centimeter), 15 centimeter above the patella with the leg in extension.
Effects of COVID-19 ARDS on ICU-AW development, ultrasonographic measurement | Change from baseline in thigh circumference at 21 days
  Using an ultrasound imaging device, the thickness of rectus femoris muscles (cm^2) were measured ultrasonographically (at the same points of anthropometric measurements) with the linear probe.
Effects of COVID-19 ARDS on ICU-AW development, scoring systems. | Change from baseline in thigh circumference at 21 days
  The muscle strength of the patients were evaluated according to the Medical Research Council (MRC) scoring.
Effects of COVID-19 ARDS on ICU-AW development, scoring systems. | Change from baseline at 21 days
  On the first day of the study, SOFA (Sequential Organ Failure Assessment) score,scoring systems were calculated for each patients.
Effects of COVID-19 ARDS on ICU-AW development, scoring systems. | Change from baseline at 21 days
  On the first day of the study, qSOFA (quick Sequential Organ Failure Assessment) score scoring systems were calculated for each patients.
Effects of COVID-19 ARDS on ICU-AW development, scoring systems. | only first day
  On the first day of the study, APACHE-II (Acute Physiology And Chronic Health Evaluation II) scoring systems were calculated for each patients.
Effects of COVID-19 ARDS on ICU-AW development, nutrition. | 21 days
  The diet of the patients were standardized by the dietitian.

CONTACTS AND LOCATIONS:
Locations (1):
- Gunes Comba Cebeci, Istanbul, Bayrampasa, Turkey (Türkiye)